CLINICAL TRIAL: NCT05217888
Title: Evaluation of Procedural Outcomes and Safety of Cerebral Embolic Protection Device for Patients Undergoing Transfemoral Transcatheter Aortic Valve Replacement in Routine Clinical Practice, A Multicenter, Prospective Observational Study
Brief Title: The Sentinel Registry
Acronym: Sentinel
Status: Completed | Type: Observational
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Professor, Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV 2022-01
Record Dates: First submitted 2022-01-17; First posted 2022-02-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Disease; Transcatheter Aortic Valve Implantation; Transcatheter Aortic Valve Replacement
Keywords: Cerebral protection
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVR: Undergoing transcatheter aortic valve replacement patients
  Interventions: Device: Sentinel

INTERVENTIONS:
Device: Sentinel — cerebral protection devices during transfemoral transcatheter aortic valve replacement

SUMMARY:
This registry is to evaluate procedural outcomes and safety outcomes of cerebral protection devices during transfemoral TAVR in real-world clinical practice.

The data from this registry will be compared with the extracted data from the TP TAVR registry(NCT038262664) using Propensity Score Matching.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Undergoing TAVR with the use of SENTINEL embolic protection device
* Higher risk of cerebrovascular embolic events (any of the followings)

  1. Bicuspid aortic valve
  2. Calcified lesion or atherosclerosis in the ascending aorta and/or aortic arch
  3. Heavy calcified aortic valve (Ca. volume > 500)
  4. Chronic kidney disease
  5. Prior stroke
  6. Stroke risk is strongly anticipated by attending physicians
* Compatible carotid and brachiocephalic artery anatomy for SENTINEL device as determined by Multi-Slice Computed Tomography scan or equivalent imaging modality
* Agrees to the study protocol and the schedule of clinical follow-up and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Vasculature in the right extremity precluding radial or brachial access
* Excessive tortuosity in the right radial/brachial/subclavian artery preventing Sentinel System access and insertion
* Inadequate circulation to the right extremity as evidenced by signs of artery occlusion (modified Allen's test) or absence of radial/brachial pulse
* Hemodialysis shunt, graft, or arterio-venous fistula involving the upper extremity vasculature
* Symptomatic or asymptomatic severe occlusive carotid disease requiring concomitant carotid endarterectomy/stenting
* Undergone carotid stenting or carotid endarterectomy within the previous 6 weeks
* Concurrent medical condition with a life expectancy of less than 1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Undergoing TAVR(transcatheter aortic valve replacement) with the use of SENTINEL embolic protection device
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
The rate of procedural success | 1 month
  Procedural Success: Sentinel system acute delivery and retrieval (categorized as successful deployment of both filters, 1 filter, or no filter and retrieval of the system)
  Procedural outcomes
  * Procedure time(min)
  * Positioning time
  * Total fluoroscopy time
  * Total contrast used
  * Total procedure index time
  * Sentinel access site vascular complications related to the procedure (major and minor)

SECONDARY OUTCOMES:
The event rate of death from any cause | 1 month
The event rate of cardiac death | 1 month
The event rate of stroke | 1 month
The event rate of myocardial infarction | 1 month
The event rate of systemic embolic event | 1 month
The event rate of vascular complication | 1 month
The event rate of bleeding | 1 month
The event rate of acute kidney injury | 1 month
The event rate of repeat hospitalization | 1 month

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Bucheon Sejong Hospital, Bucheon-si
  - Keimyung University Dongsan Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Seoul university Bundang hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung medical center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park HS, Suh CH, Ahn JM, Kang DY, Ahn SY, Wee SB, Lee SH, Seo KW, Kim MJ, Park SJ, Park DW. Effect of cerebral embolic protection device on new cerebral embolism during transcatheter aortic valve replacement: A prospective sentinel registry. Am Heart J. 2026 Jan;291:44-52. doi: 10.1016/j.ahj.2025.08.006. Epub 2025 Aug 14. PMID 40816554